CLINICAL TRIAL: NCT02405195
Title: Renal Perfusion, Filtration and Oxygenation During Cardiopulmonary Bypass (CPB)
Acronym: ECCSTUD
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lukas Lannemyr, MD, Sahlgrenska University Hospital
Other Study IDs: SahlgrenskaUHThoraxLL0
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-02

CONDITIONS: Complication of Extracorporeal Circulation; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Cardiopulmonary Bypass; Extracorporeal Circulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: cardiopulmonary bypass — During cardiac surgery, the subjects are routinely undergoing cardiopulmonary bypass
  Other Names: extracorporeal circulation

SUMMARY:
Acute kidney injury is a common complication after cardiac surgery with cardiopulmonary bypass (CPB). This study aims to investigate the effects of CPB on renal perfusion, filtration and oxygenation.

DETAILED DESCRIPTION:
After approval of the regional ethics committee, patients (n=16) undergoing combined cardiac surgery procedures during normothermic CPB will be included after informed consent. Systemic and renal variables will be measured by pulmonary artery and renal vein catheters. Glomerular filtration rate (GFR) will be measured by renal extraction of 51Cr-EDTA and renal blood flow (RBF) by the infusion clearance technique for para-aminohippuric acid (PAH) corrected for by renal extraction of PAH. Repeated measures ANOVA followed by Fisher's PLSD post-hoc test were used for statistical analyses

ELIGIBILITY:
Inclusion Criteria:

* Preserved left ventricular function (LVEF > 50%)
* Normal preoperative S-creatinine

Exclusion Criteria:

* Contraindications to radiocontrast
* Cardiac transplantation och dissection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective complex cardiac surgery
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Ricksten, Professor, Principal Investigator — Sahlgrenska Academy, dept of clinical science
Locations (1):
- Department of thoracic anesthesia, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Lannemyr L, Bragadottir G, Redfors B, Ricksten SE. Effects of milrinone on renal perfusion, filtration and oxygenation in patients with acute heart failure and low cardiac output early after cardiac surgery. J Crit Care. 2020 Jun;57:225-230. doi: 10.1016/j.jcrc.2019.12.022. Epub 2020 Jan 6. PMID 31919012

RESULTS

PARTICIPANT FLOW:
Groups:
- CardioPulmonaryBypass: Open cardiac surgery with normothermic Cardiopulmonary Bypass at 2.5 L/min/m2.
Period: Overall Study
Arm/Group | CardioPulmonaryBypass
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- CardioPulmonary Bypass: Open cardiac surgery with normothermic Cardiopulmonary Bypass at 2.5 L/min/m2.
Arm/Group | CardioPulmonary Bypass
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 18
Serum creatinine [Mean (Standard Deviation); unit: micromol per litre] | 87 (11)
Left ventricular ejection fraction [Mean (Standard Deviation); unit: %] | 58 (5)

OUTCOME MEASURES:

1. Primary Outcome: Renal Blood Flow (RBF)
Description: Renal blood flow measured with PAH clearance
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: ml per minute per 1.73 m2 body surface
Arm/Group | CardioPulmonaryBypass
Number analyzed (Participants) | 18
ml per minute per 1.73 m2 body surface
  Pre CPB | 554 (126)
  CPB 30 minutes | 524 (116)
  CPB 60 minutes | 564 (162)
  Post CPB (30 - 60 minutes) | 558 (130)
Statistical Analysis 1: Comparison: CardioPulmonaryBypass; Repeated measures ANOVA throughout measurement period (before, during and after CPB); Test type: Other; p = 0.638, ANOVA — Bonferroni-Holm adjustment for multiple comparisons was used

2. Primary Outcome: Glomerular Filtration Rate (GFR)
Description: GFR measured by renal extraction of 51Cr-EDTA
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: ml per minute per 1.73 m2 body surface
Arm/Group | CardioPulmonaryBypass
Number analyzed (Participants) | 18
ml per minute per 1.73 m2 body surface
  Before CPB | 67 (23)
  CPB 30 minutes | 68 (23)
  CPB 60 minutes | 70 (19)
  Post CPB (30 - 60 minutes) | 67 (18)
Statistical Analysis 1: Comparison: CardioPulmonaryBypass; Repeated measures ANOVA; Test type: Other; p = 0.972, ANOVA — Bonferroni-Holm adjustment for multiple comparisons was used

3. Primary Outcome: Renal Oxygenation
Description: Renal oxygen extraction, defined as renal oxygen consumption divided by renal oxygen delivery
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: fraction
Arm/Group | CardioPulmonaryBypass
Number analyzed (Participants) | 18
fraction
  Pre CPB | 0.09 (0.03)
  CPB 30 minutes | 0.12 (0.05)
  CPB 60 minutes | 0.13 (0.06)
  Post CPB (30 - 60 minutes) | 0.16 (0.05)
Statistical Analysis 1: Comparison: CardioPulmonaryBypass; Repeated measures ANOVA; Test type: Other; p < 0.001, ANOVA — Bonferroni-Holm adjustment for multiple comparisons was used

4. Secondary Outcome: Excretion of NAG
Description: Urinary biomarker of tubular renal injury
Time Frame: 24 hours
Reporting Status: Not Posted

5. Secondary Outcome: Development of Acute Kidney Injury (AKI)
Description: AKI according to AKIN criteria
Time Frame: 72 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Three days
Description: Postoperative acute kidney injury, defined as an increase in serum-creatinine ≥50 % from baseline.
Arm/Group | CardioPulmonaryBypass
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CardioPulmonaryBypass (N=18)
Acute kidney injury (Renal and urinary disorders) | 4 (4) — Increase in serum-creatinine ≥50% from baseline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No